## A Phase 3, Multicenter Study to Assess the Long Term Safety and Tolerability of ALKS 3831 in Subjects with Schizophrenia

**Unique Protocol ID:** ALK3831-A304

NCT Number: NCT02873208

**Date of Statistical Analysis** 

Plan:

11 June 2019



### STATISTICAL ANALYSIS PLAN

## ALK3831-A304 NCT02873208

Study Title: A Phase 3, Multicenter Study to Assess the Long Term Safety and

Tolerability of ALKS 3831 in Subjects with Schizophrenia

Document Status: Final Version 1.0

Document Date: 11 June 2019

Based on: ALK3831-A304 Protocol Amendment 3.0 Date: 26 Apr 2018

Sponsor: Alkermes, Inc.

852 Winter Street Waltham, MA 02451

**USA** 

#### **CONFIDENTIAL**

Information and data in this document contain trade secrets and privileged or confidential information, which is the property of Alkermes, Inc. No person is authorized to make it public without the written permission of Alkermes, Inc. These restrictions or disclosures will apply equally to all future information supplied to you that is indicated as privileged or confidential. This study is being conducted in compliance with good clinical practice, including the archiving of essential documents.

## **TABLE OF CONTENTS**

| TABLE ( | OF CONTENTS | 2 |
|---------|---------------------------------------------------------------|----|
| LIST OF | F TABLES | 4 |
| LIST OF | F FIGURES | 4 |
| ABBRE | VIATIONS | 5 |
| 1. | INTRODUCTION | 7 |
| 1.1. | Study Objectives | 7 |
| 1.1.1. | Primary Objective | 7 |
| 1.2. | Summary of the Study Design | 7 |
| 2. | SAMPLE SIZE CONSIDERATION | 8 |
| 3. | DATA ANALYSIS | 8 |
| 3.1. | General Statistical Methodology | 8 |
| 3.2. | Definitions of Analysis Populations | 9 |
| 3.2.1. | Safety Population | 9 |
| 3.2.2. | Follow-up Safety Population | 9 |
| 3.2.3. | Post-discontinuation Safety Population | 9 |
| 3.3. | Disposition | 9 |
| 3.4. | Protocol Deviation | 10 |
| 3.5. | Demographics and Baseline Characteristics | 10 |
| 3.6. | Prior and Concomitant Medication. | 10 |
| 3.7. | Treatment Adherence Rate and Extent of Exposure to Study Drug | 10 |
| 3.7.1. | Treatment Adherence Rate | 10 |
| 3.7.2. | Extent of Exposure to Study Drug. | 11 |
| 3.8. | Efficacy Analyses | 11 |
| 3.8.1. | General Considerations. | 11 |
| 3.8.2. | Efficacy Analysis | 11 |
| 3.8.3. | Other Endpoints | 12 |
| 3.8.4. | Multiple Comparison / Multiplicity | 13 |
| 3.9. | Safety Analysis | 13 |
| 3.9.1. | Adverse Events | 13 |

| 3.9.1.1. | Deaths, Serious and Other Significant AEs | 14 |
|---|---|---|
| 3.9.1.2. | Other Significant AEs. | 14 |
| 3.9.1.3. | Analysis of Abuse Potential, Withdrawal, and Dependence | 14 |
| 3.9.2. | Clinical Laboratory Parameters | 15 |
| 3.9.3. | Vital Signs, Body Weight, and ECG | 18 |
| 3.9.3.1. | Vital Signs | 18 |
| 3.9.3.2. | Weight and Body Mass Index | 19 |
| 3.9.3.3. | Electrocardiograms | 20 |
| 3.9.4. | Abnormal Movement Scales | 20 |
| 3.9.5. | Columbia-Suicide Severity Rating Scale (C-SSRS) | 21 |
| 3.10. | Pharmacokinetic/ Pharmacodynamic Data Analysis | 21 |
| 4. | INTERIM ANALYSES | 21 |
| 5. | CHANGES IN CONDUCT OR PLANNED ANALYSES FROM THE PROTOCOL | 22 |
| 6. | DEFINITIONS AND CONVENTIONS FOR HANDLING OF THE DATA | 22 |
| 6.1. | Analysis Visit Windows | 22 |
| 6.2. | Handling of Partial Dates of Concomitant Medication | 23 |
| 6.3. | Handling of Safety Data | 23 |
| 7. | GENERAL STATISTICAL METHODOLOGY | 24 |
| 7.1. | Reporting Precision | 24 |
| 8. | PROGRAMMING SPECIFICATIONS | 24 |
| 9. | MOCK TABLES, LISTINGS AND FIGURES (TLFS) | 24 |
| 10. | REFERENCES | 25 |
| APPENDI | X 1. AESI - MOVEMENT DISORDERS (INCLUDING<br>EXTRAPYRAMIDAL SYNDROME AND TARDIVE DYSKINESIA;<br>STANDARDIZED MEDDRA QUERY) | 26 |
| APPENDI | X 2. AESI - SUICIDAL IDEATION AND BEHAVIOR (CUSTOM MEDDRA QUERY) | 30 |
| APPENDI | X 3. AE TERMS - ABUSE POTENTIAL (CUSTOM MEDDRA QUERY) | 31 |
| APPENDI | X 4. AE TERMS – DEPENDENCE (CUSTOM MEDDRA QUERY) | 34 |
| APPENDI | X 5. AE TERMS – WITHDRAWAL (CUSTOM MEDRA QUERY) | 35 |

## LIST OF TABLES

| Table 1: | Definition of CGI-S Categories | 11 |
|---|---|---|
| Table 2: | Shift Categories for CGI-S response | 12 |
| Table 3: | Criteria of Potentially Clinically Significant (PCS) Abnormality for Selected Analytes | 16 |
| Table 4: | Shifts Categories from Baseline to Any Postbaseline for Selected Lipid Parameters | 17 |
| Table 5: | Shift Categories from Baseline to Any Postbaseline in Glucose and HbA1c | 18 |
| Table 6: | Shift Categories from Baseline to Any Postbaseline in Liver Function Test | 18 |
| Table 7: | Criteria for Potentially Clinically Significant (PCS) Blood Pressure or Pulse Rate | 19 |
| Table 8: | Criteria for Potentially Clinically Significant (PCS) Changes from Baseline in Body Weight | 20 |
| Table 9: | Criteria for Potentially Clinically Significant (PCS) QTcF | 20 |
| Table 10: | C-SSRS Categories for Analysis | 21 |
| Table 11: | Visit Window for All Efficacy and Safety Assessments Excluding PANSS | 22 |
| Table 12: | Visit Window for PANSS Assessments | 23 |
| Table 13: | Degree of Precision | 24 |
| | LIST OF FIGURES | |
| Figure 1: S | Study Design Schematic | 8 |

## **ABBREVIATIONS**

| Abbreviation or Term | Explanation or Definition |
|----------------------|----------------------------------------------|
| AE | Adverse event |
| AIMS | Abnormal Involuntary Movement Scale |
| BARS | Barnes Akathisia Rating Scale |
| BMI | Body mass index |
| CGI-S | Clinical Global Impression - Severity |
| C-SSRS | Columbia Suicide Severity Rating Scale |
| CMQ | Customized MedDRA queries |
| ECG | Electrocardiogram |
| eCRF | Electronic case report form |
| EPS | Extra pyramidal symptoms |
| EQ-5D | EuroQOL-5D |
| HbA1C | Hemoglobin A1c |
| IWQOL | Impact of Weight on Quality of Life |
| MedDRA | Medical Dictionary for Regulatory Activities |
| OLZ | Olanzapine |
| PANSS | Positive and Negative Syndrome Scale |
| PCS | Potentially clinically significant |
| PK | Pharmacokinetics |
| PT | Preferred term |
| KM | Kaplan-Meier |
| QTcF | QT corrected with Fridericia formula |
| SAE | Serious adverse event |
| SAP | Statistical analysis plan |
| SAS | Simpson-Angus Scale |
| SD | Standard deviation |
| SMQ | Standardized MedDRA queries |
| SOC | System organ class |
| TEAE | Treatment-emergent adverse event |

| Abbreviation or Term | Explanation or Definition |
|----------------------|---------------------------|
| ULN | Upper limit of normal |
| VAS | Visual analogue scale |
| WHO | World Health Organization |

#### 1. INTRODUCTION

This statistical analysis plan (SAP) describes the statistical methods to be used for analyses and presentation of safety and efficacy data for the study ALK3831-A304. ALK3831-A304 is a 52-week, open-label safety extension study of ALK3831-A303. This document has been prepared based on Alkermes ALK3831-A304 Study Protocol Amendment 3.0 (dated 26 April 2018)<sup>1</sup>.

#### 1.1. Study Objectives

#### 1.1.1. Primary Objective

The primary objective of this study is to evaluate the long-term safety and tolerability of ALKS 3831 in subjects with schizophrenia.

## 1.2. Summary of the Study Design

Subjects are eligible to be enrolled in the study within 7 days after completing the 24-week treatment period of the antecedent study, ALK3831-A303.

Subjects enrolled in the study will be started on the same olanzapine dose that they had maintained at the end of ALK3831-A303. Subjects taking 20 mg olanzapine (either as OLZ 20 or ALKS 3831 20/10 [20 mg olanzapine/10 mg samidorphan]) will start on ALKS 3831 20/10 in this study and subjects taking 10 mg olanzapine (either as OLZ 10 or ALKS 3831 10/10 [10 mg olanzapine/10 mg samidorphan) will start on ALKS 3831 10/10 in this study. An intermediate dose, ALKS 3831 15/10 (15 mg olanzapine/10 mg samidorphan), will also be available, and subjects may be titrated to this dose any time after the start of the study at the investigator's discretion. Dosing is flexible throughout the study; however, frequent adjustments are discouraged. Dose adjustments can only be performed on-site at the study center. Subjects requiring dose adjustments between scheduled visits should arrange an unscheduled visit for the following procedures: study drug return, adherence review, adverse event monitoring, and study drug dispensation. Safety assessments will include AE monitoring, clinical laboratory testing, vital signs, weight and waist circumference assessments, 12-lead ECGs, movement disorder assessments, including the Abnormal Involuntary Movement Scale (AIMS), Barnes Akathisia Rating Scale (BARS), Simpson Angus Scale (SAS), and the Columbia-Suicide Severity Rating Scale (C-SSRS).

Efficacy assessments to evaluate the durability of treatment effect will include Positive and Negative Syndrome Scale (PANSS) and Clinical Global Impressions-Severity (CGI-S).

Additional assessments include Impact of Weight on Quality of Life-Lite Questionnaire (IWQOL-Lite), Cigarette Use, and EuroQOL-5D (EQ-5D).

Subjects completing 52 weeks of treatment with study drug will be eligible to continue in another open-label, long-term safety study (ALK3831-A308) and will continue to receive ALKS 3831. Subjects not continuing in the ALK3831-A308 long-term safety study will enter a 4-week Safety Follow-up Period.

A schematic of the study design is provided in Figure 1.

Figure 1: Study Design Schematic



\*Visits will occur biweekly throughout the 52-week Treatment Period. Subjects will start the study on the equivalent olanzapine dose to what they maintained at the end of ALK3831-A303. The dose may be adjusted to either 10/10, 15/10, or 20/10 mg throughout the study period, based on Investigator discretion, and such dose adjustments will require subjects to visit the study site.

#### 2. SAMPLE SIZE CONSIDERATION

No formal sample size calculation is performed for this extension study. A sample size of approximately 540 is based on the estimated maximum number of subjects who might be expected to continue from the ALK3831-A303 study.

#### 3. DATA ANALYSIS

## 3.1. General Statistical Methodology

Baseline for efficacy or safety analysis is defined as the last non-missing assessment before the first dose of ALKS 3831 in the ALK3831-A304 study, and it will be used for all efficacy and safety analysis, unless specified otherwise.

Baseline of precedent study (A303) is defined as the last non-missing assessment before the first dose of study drug in the ALK3831-A303 study. It will be used for the summary of the PANSS total score and subscales and body weight results.

Treatment sequence is defined according to the treatment assignment in antecedent and current studies as ALKS 3831/ALKS 3831 (ALKS 3831 in both ALK3831-A303 study and ALK3831-A304 study) and OLZ/ALKS 3831 (olanzapine in ALK3831-A303 study and ALKS 3831 in

ALK3831-A304 study). All efficacy and safety analysis will be presented by treatment sequence and overall.

In general, descriptive statistics: n, mean, standard deviation (SD), median, minimum, and maximum, for continuous variables and number and percentage of subjects in each category for categorical variables will be provided.

All source data will be presented as subject data listings.

#### 3.2. Definitions of Analysis Populations

#### 3.2.1. Safety Population

The Safety Population will include all subjects who enrolled and received at least one dose of ALKS 3831 in the ALK3831-A304 study. All analyses will be conducted using the Safety Population except for AEs in the safety follow-up period and AE to evaluate the potential for drug withdrawal and dependence. The populations used for the analyses of these events are specified below.

#### 3.2.2. Follow-up Safety Population

Follow-up Safety Population will be defined with respect to the 5 half-lives of the product as subjects in the Safety Population and met any of the following criteria:

- Completed at least one follow-up visit after >7 days of the last dose of ALKS 3831
- Reported at least one AE reported after >7 days of the last dose of ALKS 3831

This population will be used to analyze the AEs in the safety follow-up period.

#### 3.2.3. Post-discontinuation Safety Population

Post-discontinuation Safety Population\_will be defined as subjects in the Safety Population and met any of the following criteria:

- Completed at least one follow-up visit after >2 day within 16 days of the last dose of ALKS 3831
- Reported at least one AE reported after >2 day after the last dose of ALKS 3831

AE to evaluate potential for drug withdrawal and dependence emerging following discontinuation of ALKS 3831 will be assessed for this population, during the period of >2 days to 16 days after the last dose of drug for subjects with at least 4 weeks study drug exposure.

### 3.3. Disposition

The number and percentage of subjects completing or prematurely discontinuing the study including reasons for discontinuation will be summarized for the following:

• Subjects who enrolled in the study

- Subjects in the Safety Population
- Subjects who completed the treatment period
- Subjects who discontinued treatment along with reason for discontinuation (as indicated in case report form)

#### 3.4. Protocol Deviation

Subjects with major protocol deviations in the following categories will be summarized. A supportive listing will be provided as well.

- Did not meet the study entry criteria
- Received prohibited medications
- Lack of adherence with study medication, as defined by subjects taking less than 70% of protocol specified amount of study medication
- Dosing error

#### 3.5. Demographics and Baseline Characteristics

Demographics and baseline characteristics such as sex, age, race, ethnicity, weight, and body mass index (BMI) will be summarized for the Safety Population and for the subset of subjects who participated in the patient voice substudy.

#### 3.6. Prior and Concomitant Medication

Prior medications will be defined as medications taken prior to the first dose of study drug in ALK3831-A304 study. Concomitant medications will be defined as medications taken on or after the first dose of study drug in ALK3831-A304 study. All medications will be coded using the World Health Organization WHO-DD Enhanced + Herbal (version: March 2016) or higher.

Concomitant medications taken during the treatment period will be summarized by the preferred drug name. All reported medications (including those initiated after the last dose of study medication) will be included in the listing. For the summary table, if a subject has taken a concomitant medication more than once, the subject will be counted only once for that medication.

## 3.7. Treatment Adherence Rate and Extent of Exposure to Study Drug

#### 3.7.1. Treatment Adherence Rate

Treatment adherence to the daily dosing schedule during treatment period will be summarized. Treatment adherence will be calculated as follows:

100 × Total tablets dispensed – total tablets returned – total tablets lost
Total tablets scheduled to be taken

#### 3.7.2. Extent of Exposure to Study Drug

Duration of exposure to study drug (ALKS 3831) is defined as the number of days from the date of the first dose of study drug of this study (ALK3831-A304) to the date of the last dose of study drug, inclusive (ie, last dose date – first dose date + 1 day). Duration of study drug administration will be summarized.

The overall mean and modal dose of olanzapine will be summarized

#### 3.8. Efficacy Analyses

#### 3.8.1. General Considerations

In general, continuous and categorical endpoints will be summarized using descriptive statistics based on observed data.

#### 3.8.2. Efficacy Analysis

The following endpoints will be used to evaluate durability of treatment effect:

- Change from baseline in PANSS total score, and subscales (positive, negative, and general psychopathology subscales) by visit
- Change from baseline in CGI-S by visit
- Shift analysis in CGI-S
- Time to treatment discontinuation

Summary statistics will be provided for all continuous endpoints based on observed data.

Change from current (A304) and precedent (A303) study baseline in PANSS total score and subscales will be summarized for the subset of subjects who participated in the patient voice substudy.

CGI-S response will be categorized into the categories summarized in Table 1. The number and percentage of subjects in each category and with shifts from baseline will be summarized based on the observed data by descriptive statistics at 4, 12, 24 and 52 weeks. The shift categories are summarized in Table 2.

Time to treatment discontinuation will be analyzed using the Kaplan-Meier method. Both all-cause discontinuation and discontinuation due to AE will be summarized. For prematurely discontinued subjects (all-cause or due to AE), time to discontinuation is defined as time from the date of first dose of study drug to the date of last dose of study drug. Other subjects will be censored at the last dose of the study drug.

**Table 1:** Definition of CGI-S Categories

| Response Category | CGI-S Score |
|---------------------------|-------------|
| Markedly to Extremely Ill | ≥5 |

| Response Category | CGI-S Score |
|----------------------|-------------|
| Moderately Ill | 4 |
| Normal to Mildly Ill | ≤3 |

**Table 2:** Shift Categories for CGI-S response

| Shift from Baseline Category for CGI-S Response Baseline Category Shift Category |
|---|
| Markedly to Extremely Ill |
| No change |
| ≥1 level improvement |
| 2 level improvement |
| Moderately III |
| No change |
| 1 level improvement |
| 1 level worsening |
| Normal to Mildly Ill |
| No change |
| ≥1 level worsening |
| 2 level worsening |

#### 3.8.3. Other Endpoints

- Change from baseline in IWQOL-Lite scales (total score, physical function, self-esteem, sexual life, public distress, and work) by visit
- Change from baseline in EQ-5D-5L index value and visual analogue scale (VAS) score by visit

Descriptive statistics of IWQOL-Lite scales and EQ-5D-5L, including n, mean, SD, median, minimum, and maximum, will be summarized by visit based on observed data.

The IWQOL-Lite scale is a 31-item self-report measure of obesity-specific quality of life. IWQOL-Lite provides an overall total score as well as scores on five domains: (1) physical function, (2) self-esteem, (3) sexual life, (4) public distress, and (5) work. The raw scores will be transformed as follows (Tessier et al, 2012)<sup>3</sup>: the transformed scores range from 0 to 100, with 100 representing the best, and 0 representing the most impaired quality of life.

$$Transformed\ Score = \frac{maximum\ theoretical\ score - actual\ score}{test\ score\ range} X100$$

The EQ-5D-5L is a validated quality of life questionnaire developed by the EuroQol Group in order to provide a simple, generic utility measure for characterizing current health states of patients. EQ-5D-5L is designed for self-completion by subjects. It consists of 2 parts – the EQ-5D-5L descriptive system and the VAS.

The EQ-5D-5L descriptive system comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels.

The 5 dimensional 5-level systems are converted into an index value. Values for theoretically possible health states are calculated using a regression model and weighted according to the social preferences of the U.S. population (Van Hout et al, 2012)<sup>4</sup>. The VAS records the respondent's self-rated health on a vertical VAS. The VAS has 100 (Best health you can imagine) at the top, and 0 (Worst health you can imagine) at the bottom. This information can be used as a quantitative measure of health outcomes as judged by the individual respondents. EQ-5D-5L self-reported VAS data generates information on the self-perceived overall health-related quality of life. Change from baseline in EQ-5D-5L index value and VAS score will be analyzed.

#### 3.8.4. Multiple Comparison / Multiplicity

Not applicable.

#### 3.9. Safety Analysis

#### 3.9.1. Adverse Events

Incidence of treatment emergent AEs (TEAEs) will be analyzed as a safety endpoint. Adverse events will be coded by System Organ Class and Preferred Term using the Medical Dictionary for Regulatory Activities (MedDRA®) Version 21.0 or higher. The verbatim term will be included in the AE listings.

An AE (coded by preferred term) will be considered as a TEAE if the event is newly occurring or worsening on or after the date of first dose of study drug and within 7 days after the last dose of study drug in this study.

An overview table, including number of subjects with TEAEs, AEs leading to treatment discontinuation, study drug related TEAEs, and SAEs will be provided.

The incidence (number and percentage) of subjects reporting TEAEs during the treatment period will be presented for the following categories:

- System organ class and preferred term
- Preferred term, and including the following subset:
  - TEAEs experienced by ≥2% of subjects (in any group)
- System organ class, preferred term, and severity
- System organ class, preferred term for severe TEAEs

- System organ class, preferred term, and relationship
- System organ class, preferred term for study drug related TEAEs

If the same preferred term occurred more than once for the same subject, the subject will be counted only once for that preferred term using the most severe and most related occurrence for the summarization by severity and by relationship to the study drug.

In addition, the number and percentage of subjects reporting AEs during the safety follow-up period will be tabulated by the system organ class and preferred term.

Subgroup analysis by age (<40 years vs ≥40 years), sex (Female vs Male) and race (Black or African American, White, and Other) will be performed for TEAEs during the treatment period by preferred term.

#### 3.9.1.1. Deaths, Serious and Other Significant AEs

The number and percentage of subjects who have serious adverse events (SAEs) and AEs leading to premature discontinuation from the treatment will be summarized by system organ class and preferred term.

By-subject listings will be provided for SAEs, AEs leading to treatment discontinuation and AEs leading to death.

#### 3.9.1.2. Other Significant AEs

In addition, incidence of a selected subset of relevant AEs in this class of drugs (e.g., Extrapyramidal symptoms [EPS) TEAEs, TEAE to evaluate potential of suicidal ideation and behavior, etc.) will be summarized by preferred term. The selection of AEs per subset will be based on the preferred terms from Standardized MedDRA queries (SMQs) or Customized MedDRA queries (CMQ's).

#### 3.9.1.3. Analysis of Abuse Potential, Withdrawal, and Dependence

#### 3.9.1.3.1. Analysis of Abuse Potential

Number and percentage subjects with TEAEs to evaluate abuse potential will be summarized by category (abuse behavior, euphoria related, and non-specific) and preferred term. The selection of AEs per subset will be based on the preferred terms from Customized MedDRA queries (CMQs).

#### 3.9.1.3.2. Analysis of Withdrawal and Dependence

Adverse events with an onset date within 2 weeks (>2 to  $\leq$ 16 days) after the last dose of the study drug in those subjects who have received at least 4 weeks of study drug will be included in the evaluation of the potential for withdrawal and dependence. The selection of AEs per subset will be based on the preferred terms from Customized MedDRA queries (CMQs).

The number and percentage of subjects with such AEs will be summarized in the Post-discontinuation Safety Populations by preferred term for subjects with a duration of study drug exposure ≥4 weeks.

#### 3.9.2. Clinical Laboratory Parameters

Laboratory parameters will be presented in conventional (ie, US) units. Only scheduled laboratory parameters will be included in the summaries, unless specified otherwise. All laboratory data, including those collected at unscheduled visits, will be included in the listings.

Laboratory results including baseline and change from baseline during the treatment period for chemistry and hematology parameters will be summarized by visit.

Clinical laboratory test values, scheduled or unscheduled, will be considered potentially clinically significant (PCS) if they meet PCS criteria listed in Table 3. The number and percentage of subjects who have postbaseline PCS clinical laboratory values will be summarized. The percentages will be calculated based on the number of subjects with non-PCS baseline value and have at least one postbaseline assessment. All PCS values including baseline PCS values will be included in supportive listings.

For selected metabolic parameters (fasting total cholesterol, fasting high density lipoprotein[HDL], fasting low density lipoprotein[LDL], fasting triglycerides, fasting glucose, and hemoglobin A1c[HbA1c]), an analysis of sustained PCS values will also be conducted. The percentage of subjects with sustained PCS values through the treatment period will be summarized. The denominator is all subjects with non-PCS at baseline and at least two postbaseline assessments, and the numerator is the number of subjects who met PCS criteria at the last 2 assessments within the treatment period.

Shift tables for selected fasting metabolic parameters (total cholesterol, LDL, HDL, triglycerides, glucose and HbA1c) and liver function tests will be presented. The criteria are summarized in Table 4, Table 5 and Table 6.

Table 3: Criteria of Potentially Clinically Significant (PCS) Abnormality for Selected Analytes

| Parameter | Criteria |
|-----------------------------------|-------------------------------|
| Chemistry | |
| Albumin | <2.5 g/dL |
| Alkaline Phosphatase (U/L) | ≥3 × ULN |
| Alanine Aminotransferase (U/L) | ≥3 × ULN |
| Aspartate Aminotransferase (U/L) | ≥3 × ULN |
| Bilirubin, Total | ≥2.0 mg/dL |
| Blood Urea Nitrogen | >30 mg/dL |
| Cholesterol, Random | >300 mg/dL |
| Cholesterol, Fasting <sup>a</sup> | ≥240 mg/dL |
| Cholesterol, Fasting | Increase ≥40 mg/dL |
| Cholesterol, HDL Fasting | <40 mg/dL |
| Cholesterol, HDL Fasting | Decrease ≥20 mg/dL |
| Cholesterol, LDL Fasting | ≥160 mg/dL |
| Cholesterol, LDL Fasting | Increase ≥30 mg/dL |
| Creatine Kinase (U/L) | ≥3 × ULN |
| Creatinine | ≥2.0 mg/dL |
| Glucose, Random | <50 mg/dL or<br>≥200 mg/dL |
| Glucose, Fasting | <50 mg/dL or<br>≥126 mg/dL |
| Glucose, Fasting | Increase ≥10 mg/dL |
| HbA1c | ≥ 5.7% |
| Potassium | <3 mmol/L or<br>>5.5 mmol/L |
| Lactate Dehydrogenase (U/L) | >3 × ULN |
| Prolactin (Female) | >30 ng/mL |
| Prolactin (Male) | >20 ng/mL |
| Sodium | <130 mmol/L or<br>>150 mmol/L |

Table 3: Criteria of Potentially Clinically Significant (PCS) Abnormality for Selected Analytes (Continued)

| Triglycerides, Fasting | ≥200 mg/dL |
|---|---|
| Triglycerides, Fasting | Increase ≥50 mg/dL |
| Hematology | |
| Eosinophils | $>1.0 \times 10^3/\mu$ L |
| Hematocrit (Female) | ≤32% |
| Hematocrit (Male) | ≤37% |
| Neutrophils, Absolute | $<1.5 \times 10^3/\mu$ L |
| Platelets | $<75.0 \times 10^3 \text{ cells/}\mu\text{L or}$<br>$\geq 700.0 \times 10^3 \text{ cells/}\mu\text{L}$ |
| Leukocytes | $\leq 2.8 \times 10^{3}/\mu L \text{ or}$<br>$\geq 16.0 \times 10^{3}/\mu L$ |

<sup>&</sup>lt;sup>a</sup> reported fasting.

Table 4: Shifts Categories from Baseline to Any Postbaseline for Selected Lipid Parameters

| Total Cholesterol (fasting) mg/dL |
|---------------------------------------------|
| Normal (<200) to High (≥240) |
| Borderline (≥200 and < 240) to High (≥240) |
| Normal (<200) to Borderline (≥200 and <240) |
| LDL Cholesterol (fasting) mg/dL |
| Normal (<100) to High (≥160) |
| Borderline (≥100 and <160) to High (≥160) |
| Normal (<100) to Borderline (≥100 and <160) |
| HDL Cholesterol (fasting) mg/dL |
| Normal (≥40) to Low (<40) |
| Triglycerides (fasting) mg/dL |
| Normal (<150) to High (≥200) |
| Borderline (≥150 and <200) to High (≥200) |
| Normal (<150) to Borderline (≥150 and <200) |

#### Table 5: Shift Categories from Baseline to Any Postbaseline in Glucose and HbA1c

| Glucose (fasting) mg/dL |
|------------------------------------------------|
| Normal (<100) to Impaired (≥100 and <126) |
| Normal (<100) to High (≥126) |
| Impaired (≥100 and <126) to High (≥126) |
| HbA1c % |
| Normal (<5.7%) to Borderline (≥5.7% and <6.5%) |
| Borderline (≥5.7% and <6.5%) to High (≥6.5%) |
| Normal (<5.7%) to High (≥6.5%) |

#### Table 6: Shift Categories from Baseline to Any Postbaseline in Liver Function Test

| Alanine Aminotransferase (ALT) (U/L) |
|----------------------------------------|
| Shift from Normal to ≥3 x ULN |
| Shift from Normal to ≥5 x ULN |
| Shift from Normal to ≥10 x ULN |
| Aspartate Aminotransferase (AST) (U/L) |
| Shift from Normal to ≥3 x ULN |
| Shift from Normal to ≥5 x ULN |
| Shift from Normal to ≥10 x ULN |
| Bilirubin, Total (mg/dL) |
| Shift from Normal to >1 x ULN |
| Shift from Normal to ≥2 x ULN |

#### 3.9.3. Vital Signs, Body Weight, and ECG

#### **3.9.3.1.** Vital Signs

Descriptive statistics for vital signs and changes from baseline values at each scheduled time point will be presented.

Vital sign values will be considered PCS if they meet both the observed-value criteria and the change-from-baseline criteria listed in Table 7. The number and percentage of subjects with PCS postbaseline values will be tabulated. The percentages will be calculated based on the number of subjects with non-PCS baseline values and at least one postbaseline assessment. The numerator

will be the number of subjects with non-PCS baseline values and at least one postbaseline PCS value. A supportive listing of subjects with PCS postbaseline values will be provided.

All vital signs will be presented in the subject data listing.

Orthostatic hypotension (20/10 mmHg) is defined as a fall in systolic blood pressure of at least 20 mmHg and a fall in the diastolic blood pressure of at least 10 mmHg upon standing from supine. Orthostatic hypotension (30 mmHg) is defined as a fall in systolic blood pressure of at least 30 mmHg upon standing from supine.

Orthostatic tachycardia is defined as a heart rate increase of 30 beats per minute (bpm) or more upon standing from supine, or over 120 bpm upon standing.

The number and percentage of subjects with orthostatic hypotension or orthostatic tachycardia occurring at any postbaseline visit will be summarized.

Table 7: Criteria for Potentially Clinically Significant (PCS) Blood Pressure or Pulse Rate

| Parameter | Criteria |
|---|---|
| Supine Systolic Blood Pressure | ≤90 and decrease ≥20 mm Hg<br>≥180 and increase ≥20 mm Hg |
| Supine Diastolic Blood Pressure | ≤50 and decrease ≥15 mm Hg<br>≥105 and increase ≥15 mm Hg |
| Supine Heart Rate | ≤50 and decrease ≥15 bpm<br>≥120 and increase ≥15 bpm |

#### 3.9.3.2. Weight and Body Mass Index

Body weight (kg), BMI (kg/m²) and waist circumferences (cm) (baseline and change from baseline) will be summarized using observed data. Absolute (kg) and percent change from baseline in body weight will be summarized by visit.

Absolute and percent change from current (A304) and precedent (A303) study baseline in body weight will also be summarized for the subset of subjects who participated in the patient voice substudy.

Number and percentage of subjects with  $\geq$ 7% or  $\geq$ 10% weight gain from baseline based on the observed data will be summarized by visit. In addition, number and percentage of subjects with weight change values considered as PCS occurring at any postbaseline visit will be summarized. Criteria for PCS are presented below. The percentages will be calculated relative to the number of subjects in the Safety Population with at least one postbaseline value. A supportive listing will be provided for subjects with PCS values.

Table 8: Criteria for Potentially Clinically Significant (PCS) Changes from Baseline in Body Weight

| Parameter | Criteria |
|-------------|----------------------------|
| Body Weight | Decrease from Baseline ≥7% |
| | Increase from Baseline ≥7% |

#### 3.9.3.3. Electrocardiograms

Descriptive statistics for ECG parameters (heart rate, PR interval, RR interval, QRS interval, QT interval, and QTc interval) at baseline and change from baseline values at each scheduled assessment timepoint and at the end of the treatment period will be presented. QTc interval will be calculated using Fridericia (QTcF = QT/(RR) $^{1/3}$ ) corrections; if RR is not available, it will be replaced with 60/HR in the correction formula.

Electrocardiogram parameter values are considered PCS if they meet or exceed the higher-limit PCS criteria listed in Table 9. The number and percentage of subjects with PCS postbaseline ECG values will be tabulated. The percentages will be calculated based on the number of subjects with non-PCS baseline values and at least one postbaseline assessment. The numerator is the number of subjects with non-PCS baseline values and at least one postbaseline PCS value. A supportive listing of subjects with PCS values will be provided.

Table 9: Criteria for Potentially Clinically Significant (PCS) QTcF

| Parameter | Criteria |
|-----------|--------------------------------------|
| QTcF | >450 to ≤480 msec |
| | >480 to ≤500 msec |
| | >500 msec |
| | Change from baseline >30 to ≤60 msec |
| | Change from baseline >60 msec |

#### 3.9.4. Abnormal Movement Scales

Extra pyramidal symptoms (EPS) will be evaluated as AEs and also as assessed by abnormal movement scales. Abnormal movement scales will include the following: Abnormal Involuntary Movement Scale (AIMS), Barnes Akathisia Rating Scale (BARS), and Simpson-Angus Scale (SAS).

Change from baseline in all abnormal movement scales, total scores and subscale scores will be summarized by visit.

Number and percentage of subjects meeting the criteria for treatment emergent Parkinsonism (SAS total score>3), for treatment emergent akathisia (BARS global clinical assessment of akathisia score ≥2), for treatment emergent dyskinesia (AIMS score ≥3 on any of the first

7 items, or a score  $\geq 2$  on two or more of any of the first 7 items) at any postbaseline visit will be summarized.

A listing will be provided for every abnormal movement scale. Listing for treatment emergent EPS will be provided.

#### 3.9.5. Columbia-Suicide Severity Rating Scale (C-SSRS)

The C-SSRS is a questionnaire used to measure the presence and intensity of suicidal ideation and behavior. Suicidal behavior and suicidal ideation will be summarized descriptively (Table 10). The number of subjects with suicidal ideation and suicidal behavior will be summarized.

Supportive tabular display of subjects with all values will be provided.

**Table 10:** C-SSRS Categories for Analysis

| Category | C-SSRS Item response is "YES" |
|---|---|
| Suicidal behavior <sup>a</sup> | Preparatory acts or behavior |
| | Aborted attempt |
| | Interrupted attempt |
| | Actual attempt |
| | Complete suicide |
| Suicidal ideation <sup>a</sup> | Wish to be dead |
| | Non-specific active suicidal thoughts |
| | Active suicidal ideation with any methods (not plan) without intent to act |
| | Active suicidal ideation with some intent to act, without specific |
| | plan |
| | Active suicidal ideation with specific plan and intent |
| Non-Suicidal Self-Injurious | Non-Suicidal Self-Injurious |
| Behavior | Behavior |

<sup>&</sup>lt;sup>a</sup> Derived based on responses to individual items listed within the category

### 3.10. Pharmacokinetic/ Pharmacodynamic Data Analysis

Not applicable.

#### 4. INTERIM ANALYSES

No interim analysis is planned for this study.

## 5. CHANGES IN CONDUCT OR PLANNED ANALYSES FROM THE PROTOCOL

To further assess the long-term durability, the following analysis was added in SAP but were not specified in protocol.

• Shift analysis in CGI-S

## 6. DEFINITIONS AND CONVENTIONS FOR HANDLING OF THE DATA

Dataset specifications will be provided in a separate document.

#### 6.1. Analysis Visit Windows

Scheduled analysis visits are visits at scheduled timepoints as specified in the protocol (Table 3 Schedule of Visits and Assessments).

Scheduled analysis visits during the study period will be the same as the nominal visits collected in eCRF. There will be one valid value of assessment kept for each scheduled analysis visit in summary/analysis statistics.

Unscheduled visits are visits with data not collected on the scheduled time point. Unscheduled visits will not be used for by-visit summary/analysis statistics, unless specified otherwise.

All unscheduled visits as collected in eCRF will be included in listings.

Last postbaseline values are defined as the last valid postbaseline values collected for each subject during the treatment period.

An early termination (ET) visit during the on-treatment period can be mapped to a scheduled visit, if there is no valid value already at that visit. Visit windows are defined in Table 11 and Table 12. An ET visit that is not mapped will not be summarized in the tables or figures, but will be included in the listing.

Table 11: Visit Window for All Efficacy and Safety Assessments Excluding PANSS

| Analysis Visit to be<br>Mapped to | Target Study Week | Target Visit Day <sup>a</sup> | Visit Window |
|---|---|---|---|
| Visit 1 | Week 0 | Day 1 | 1 |
| Visit 2 | Week 2 | Day 15 | [2, 21] |
| Visit 3 | Week 4 | Day 29 | [22, 35] |
| Visit 4 | Week 6 | Day 43 | [36, 49] |
| Visit 5 | Week 8 | Day 57 | [50, 70] |
| Visit 7 | Week 12 | Day 85 | [71, 98] |

| Analysis Visit to be<br>Mapped to | Target Study Week | Target Visit Day <sup>a</sup> | Visit Window |
|---|---|---|---|
| Visit 9 | Week 16 | Day 113 | [99, 126] |
| Visit 11 | Week 20 | Day 141 | [127, 154] |
| Visit 13 | Week 24 | Day 169 | [155, 182] |
| Visit 15 | Week 28 | Day 197 | [183, 210] |
| Visit 17 | Week 32 | Day 225 | [211, 238] |
| Visit 19 | Week 36 | Day 253 | [239, 266] |
| Visit 21 | Week 40 | Day 281 | [267, 294] |
| Visit 23 | Week 44 | Day 309 | [295, 322] |
| Visit 25 | Week 48 | Day 337 | [323, 350] |
| Visit 27 | Week 52 | Day 365 | [351, 371] |

<sup>&</sup>lt;sup>a</sup> Visit Day is calculated as date of visit – date of the first dose of study drug + 1 day.

**Table 12: Visit Window for PANSS Assessments** 

| Analysis Visit to be<br>Mapped to | Target Study Week | Target Visit Day | Visit Window |
|---|---|---|---|
| Visit 2 | Week 2 | Day 15 | [2, 21] |
| Visit 3 | Week 4 | Day 29 | [22, 42] |
| Visit 5 | Week 8 | Day 57 | [43, 70] |
| Visit 7 | Week 12 | Day 85 | [71, 126] |
| Visit 13 | Week 24 | Day 169 | [127, 210] |
| Visit 19 | Week 36 | Day 253 | [211, 308] |
| Visit 27 | Week 52 | Day 365 | [309, 371] |

## **6.2.** Handling of Partial Dates of Concomitant Medication

Partial start dates of prior and concomitant medications will be assumed to be the earliest possible date consistent with the partial date. Partial stop dates of prior and concomitant medications will be assumed to be the latest possible date consistent with the partial date. In the case of completely missing stop date, medication will be assumed to be ongoing.

## 6.3. Handling of Safety Data

All efforts should be made to obtain the missing information from the investigator. For C-SSRS, vital signs, laboratory testing (chemistry, hematology, urinalysis), and 12-lead ECGs, only observed data will be used for analyses, and missing data will not be imputed.

#### 7. GENERAL STATISTICAL METHODOLOGY

In general, summary statistics (n, mean, SD, median, minimum, and maximum for continuous variables, and number and percentage of subjects in each category for categorical variables) will be provided by treatment sequence and overall. All summary tables will be based on observed data, and missing values will not be imputed. Measurements collected from unscheduled visits or repeated assessments will not be included in the by-visit summary tables or figures, but will be included in the analyses for the PCS postbaseline values, and subject listings. Source data for the summary tables will be presented as subject data listings.

### 7.1. Reporting Precision

Summary statistics will be presented to the following degree of precision, unless otherwise specified:

**Table 13:** Degree of Precision

| Statistics | Degree of Precision |
|---|---|
| Mean, Median, Confidence limit boundaries | One more than the raw data, up to 3 decimal places. |
| Standard deviation, Standard error | One more than the mean, up to 3 decimal places |
| Minimum, Maximum | The same as the raw data, up to 2 decimal places |
| P-value | Rounded to 3 decimal places and therefore presented as 0.xxx; <i>P</i> -values smaller than 0.001 as '<0.001'; P-values greater than 0.999 as '>0.999'. |
| Percentage | One decimal place. A percentage of 100% will be reported as 100%. Percentages of zero will be reported as 0. |

Fractional numeric values will be presented with a zero to the left of the decimal point (for example, 0.12 - 0.30).

For weight, height, and BMI, one decimal place will be used for summary statistics, unless otherwise specified.

#### 8. PROGRAMMING SPECIFICATIONS

Programming specifications will be provided in a separate document.

### 9. MOCK TABLES, LISTINGS AND FIGURES (TLFS)

Mock-up tables and listings will be provided in a separate document.

#### 10. REFERENCES

- 1. Alkermes ALK3831-A304 Study Protocol Amendment 3.0 Date: 26 April 2018
- 2. Marder SR, Davis JM, Chouinard G. The effects of risperidone on the five dimensions of schizophrenia derived by factor analysis: combined results of the North American trials. *J Clin Psychiatry*. 1997; 58(12): 538-546.
- 3. Tessier A et al. Understanding the Determinants of Weight-Related Quality of Life among Bariatric Surgery Candidates. *Journal of Obesity* 2012; 2012: 713426
- 4. Van Hout B, Janssen MF, et al. Interim scoring for the EQ-5D-5L: Mapping the EQ-5D-5L to EQ-5D-3L value sets. *Value in Health* 2012 Jul-Aug;15(5):708-15

# APPENDIX 1. AESI - MOVEMENT DISORDERS (INCLUDING EXTRAPYRAMIDAL SYNDROME AND TARDIVE DYSKINESIA; STANDARDIZED MEDDRA QUERY)

| Preferred Term (SMQ [#20000095] of Extrapyramidal syndrome) | PT Code |
|-------------------------------------------------------------|----------|
| Abnormal involuntary movement scale | 10075002 |
| Action tremor | 10072413 |
| Akathisia | 10001540 |
| Akinesia | 10001541 |
| Athetosis | 10003620 |
| Ballismus | 10058504 |
| Blepharospasm | 10005159 |
| Bradykinesia | 10006100 |
| Bradyphrenia | 10050012 |
| Buccoglossal syndrome | 10006532 |
| Chorea | 10008748 |
| Choreoathetosis | 10008754 |
| Chronic tic disorder | 10076661 |
| Cogwheel rigidity | 10009848 |
| Complex tic | 10076663 |
| Dopamine dysregulation syndrome | 10067468 |
| Dopa-responsive dystonia | 10080034 |
| Drooling | 10013642 |
| Dyskinesia | 10013916 |
| Dyskinesia neonatal | 10013922 |
| Dyskinesia oesophageal | 10013924 |
| Dysphonia | 10013952 |
| Dystonia | 10013983 |
| Dystonic tremor | 10073210 |
| Early onset primary dystonia | 10076668 |
| Emprosthotonus | 10014566 |
| Extrapyramidal disorder | 10015832 |

| Preferred Term (SMQ [#20000095] of Extrapyramidal syndrome) | PT Code |
|-------------------------------------------------------------|----------|
| Facial spasm | 10063006 |
| Fine motor skill dysfunction | 10076288 |
| Freezing phenomenon | 10060904 |
| Gait disturbance | 10017577 |
| Gait inability | 10017581 |
| Grimacing | 10061991 |
| Hyperkinesia | 10020651 |
| Hyperkinesia neonatal | 10020652 |
| Hypertonia | 10020852 |
| Hypertonia neonatal | 10048615 |
| Hypokinesia | 10021021 |
| Hypokinesia neonatal | 10021022 |
| Laryngeal tremor | 10078751 |
| Laryngospasm | 10023891 |
| Meige's syndrome | 10027138 |
| Micrographia | 10057333 |
| Mobility decreased | 10048334 |
| Motor dysfunction | 10061296 |
| Movement disorder | 10028035 |
| Muscle contractions involuntary | 10028293 |
| Muscle rigidity | 10028330 |
| Muscle spasms | 10028334 |
| Muscle spasticity | 10028335 |
| Muscle tightness | 10049816 |
| Muscle tone disorder | 10072889 |
| Muscle twitching | 10028347 |
| Musculoskeletal stiffness | 10052904 |
| Oculogyric crisis | 10030071 |
| Oesophageal spasm | 10030184 |
| On and off phenomenon | 10030312 |

| Preferred Term (SMQ [#20000095] of Extrapyramidal syndrome) | PT Code |
|-------------------------------------------------------------|----------|
| Opisthotonus | 10030899 |
| Oromandibular dystonia | 10067954 |
| Oropharyngeal spasm | 10031111 |
| Parkinsonian crisis | 10048868 |
| Parkinsonian gait | 10056242 |
| Parkinsonian rest tremor | 10056437 |
| Parkinsonism | 10034010 |
| Parkinsonism hyperpyrexia syndrome | 10071243 |
| Parkinson's disease | 10061536 |
| Parkinson's disease psychosis | 10074835 |
| Pharyngeal dyskinesia | 10070912 |
| Pleurothotonus | 10035628 |
| Postural reflex impairment | 10067206 |
| Postural tremor | 10073211 |
| Posture abnormal | 10036436 |
| Posturing | 10036437 |
| Protrusion tongue | 10037076 |
| Provisional tic disorder | 10076694 |
| Psychomotor hyperactivity | 10037211 |
| Rabbit syndrome | 10068395 |
| Reduced facial expression | 10078576 |
| Respiratory dyskinesia | 10057570 |
| Resting tremor | 10071390 |
| Restlessness | 10038743 |
| Risus sardonicus | 10039198 |
| Secondary tic | 10076702 |
| Spasmodic dysphonia | 10067672 |
| Tardive dyskinesia | 10043118 |
| Tic | 10043833 |
| Tongue spasm | 10043981 |

| Preferred Term (SMQ [#20000095] of Extrapyramidal syndrome) | PT Code |
|-------------------------------------------------------------|----------|
| Torticollis | 10044074 |
| Torticollis psychogenic | 10044076 |
| Tremor | 10044565 |
| Tremor neonatal | 10044575 |
| Trismus | 10044684 |
| Uvular spasm | 10050908 |
| Walking disability | 10053204 |
| Writer's cramp | 10072249 |

## APPENDIX 2. AESI - SUICIDAL IDEATION AND BEHAVIOR (CUSTOM MedDRA QUERY)

| Preferred Term | PT Code |
|-------------------------------------------------|----------|
| Columbia suicide severity rating scale abnormal | 10075616 |
| Completed suicide | 10010144 |
| Depression suicidal | 10012397 |
| Intentional overdose | 10022523 |
| Intentional self-injury | 10022524 |
| Overdose | 10033295 |
| Poisoning deliberate | 10036000 |
| Self-injurious ideation | 10051154 |
| Suicidal behaviour | 10065604 |
| Suicidal ideation | 10042458 |
| Suicide attempt | 10042464 |
| Suicide threat | 10077417 |

## APPENDIX 3. AE TERMS - ABUSE POTENTIAL (CUSTOM MedDRA QUERY)

| Category | Preferred Term | PT Code |
|----------------|-----------------------------------------------|----------|
| Abuse behavior | Accidental overdose | 10000381 |
| | Drug abuse | 10013654 |
| | Drug abuser | 10061111 |
| | Drug detoxification | 10052237 |
| | Drug diversion | 10066053 |
| | Drug level above therapeutic | 10061132 |
| | Drug level increased | 10013722 |
| | Drug screen | 10050837 |
| | Drug screen positive | 10049177 |
| | Drug use disorder | 10079381 |
| | Drug use disorder, antepartum | 10079382 |
| | Drug use disorder, postpartum | 10079383 |
| | Intentional overdose | 10022523 |
| | Intentional product misuse | 10074903 |
| | Intentional product use issue | 10076308 |
| | Maternal use of illicit drugs | 10026938 |
| | Needle track marks | 10028896 |
| | Neonatal complications of substance abuse | 10061862 |
| | Overdose | 10033295 |
| | Prescription drug used without a prescription | 10076639 |
| | Prescription form tampering | 10067669 |
| | Product tampering | 10069330 |
| | Reversal of opiate activity | 10039004 |
| | Substance abuse | 10066169 |
| | Substance abuser | 10067688 |
| | Substance use | 10070964 |
| | Substance use disorder | 10079384 |
| | Substance-induced mood disorder | 10072387 |

| Category | Preferred Term | PT Code |
|------------------|------------------------------------------|----------|
| | Substance-induced psychotic disorder | 10072388 |
| | Toxicity to various agents | 10070863 |
| Euphoria related | Euphoric mood | 10015535 |
| | Feeling abnormal | 10016322 |
| | Feeling drunk | 10016330 |
| | Feeling of relaxation | 10016352 |
| | Hallucination | 10019063 |
| | Hallucination, auditory | 10019070 |
| | Hallucination, gustatory | 10019071 |
| | Hallucination, olfactory | 10019072 |
| | Hallucination, synaesthetic | 10062824 |
| | Hallucination, tactile | 10019074 |
| | Hallucination, visual | 10019075 |
| | Hallucinations, mixed | 10019079 |
| | Inappropriate affect | 10021588 |
| | Mood altered | 10027940 |
| | Mood swings | 10027951 |
| | Thinking abnormal | 10043431 |
| Non-specific | Acute psychosis | 10001022 |
| | Aggression | 10001488 |
| | Cognitive disorder | 10057668 |
| | Confusional state | 10010305 |
| | Delirium | 10012218 |
| | Delusional disorder, unspecified type | 10012255 |
| | Depersonalisation/derealisation disorder | 10077805 |
| | Disorientation | 10013395 |
| | Dissociation | 10013457 |
| | Disturbance in attention | 10013496 |
| | Disturbance in social behaviour | 10061108 |
| | Dizziness | 10013573 |

| Category | Preferred Term | PT Code |
|----------|---------------------------------|----------|
| | Dopamine dysregulation syndrome | 10067468 |
| | Emotional disorder | 10014551 |
| | Flight of ideas | 10016777 |
| | Medication overuse headache | 10072720 |
| | Mental impairment | 10027374 |
| | Narcotic bowel syndrome | 10072286 |
| | Paranoia | 10033864 |
| | Psychotic behaviour | 10037249 |
| | Psychotic disorder | 10061920 |
| | Sedation | 10039897 |
| | Somnolence | 10041349 |
| | Stupor | 10042264 |

## APPENDIX 4. AE TERMS – DEPENDENCE (CUSTOM MedDRA QUERY)

| Preferred Term | PT Code |
|-----------------------------|----------|
| Dependence | 10012335 |
| Drug dependence | 10013663 |
| Drug dependence, antepartum | 10013675 |
| Drug dependence, postpartum | 10013676 |
| Drug tolerance | 10052804 |
| Drug tolerance decreased | 10052805 |
| Drug tolerance increased | 10052806 |
| Substance dependence | 10076595 |

## APPENDIX 5. AE TERMS – WITHDRAWAL (CUSTOM MedRA QUERY)

| Preferred Term | PT Code |
|-------------------------------------|----------|
| Abdominal pain | 10000081 |
| Agitation | 10001497 |
| Anhedonia | 10002511 |
| Anxiety | 10002855 |
| Arthralgia | 10003239 |
| Chills | 10008531 |
| Depressed mood | 10012374 |
| Depression | 10012378 |
| Diarrhoea | 10012735 |
| Drug detoxification | 10052237 |
| Drug rehabilitation | 10064773 |
| Drug withdrawal convulsions | 10013752 |
| Drug withdrawal headache | 10013753 |
| Drug withdrawal maintenance therapy | 10052970 |
| Drug withdrawal syndrome | 10013754 |
| Drug withdrawal syndrome neonatal | 10013756 |
| Dysphoria | 10013954 |
| Dyssomnia | 10061827 |
| Feeling of despair | 10016344 |
| Headache | 10019211 |
| Hyperhidrosis | 10020642 |
| Insomnia | 10022437 |
| Irritability | 10022998 |
| Morose | 10027977 |
| Mydriasis | 10028521 |
| Nausea | 10028813 |
| Negative thoughts | 10058672 |
| Nervousness | 10029216 |

| Preferred Term | PT Code |
|--------------------------------|----------|
| Obsessive thoughts | 10029897 |
| Pain | 10033371 |
| Persistent depressive disorder | 10077804 |
| Piloerection | 10035039 |
| Poor quality sleep | 10062519 |
| Rebound effect | 10038001 |
| Restlessness | 10038743 |
| Reversal of opiate activity | 10039004 |
| Rhinorrhoea | 10039101 |
| Steroid withdrawal syndrome | 10042028 |
| Syncope | 10042772 |
| Tachycardia | 10043071 |
| Terminal insomnia | 10068932 |
| Tremor | 10044565 |
| Vomiting | 10047700 |
| Withdrawal arrhythmia | 10047997 |
| Withdrawal syndrome | 10048010 |
| Yawning | 10048232 |